CLINICAL TRIAL: NCT01399567
Title: Nursing Home Pain Management Algorithm Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Responsible Party: Mary Ersek PhD, RN, University of Pennsylvania School of Nursing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5R01NR009100 (NIH)
Record Dates: First submitted 2011-06-23; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Pain
Keywords: pain; depression; nursing homes; diffusion of innovations; clinical trial
MeSH Terms: conditions — Pain; Depression | interventions — Algorithms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Algorithm (Experimental): The NH pain management algorithm is a series of decision-making tools that begins with regular, comprehensive pain assessment matched to residents' cognitive status and proceed through analgesic therapy appropriate to the character, severity, and pattern of pain. The algorithm is coupled with intense diffusion strategies (e.g., education, consultation, boosters) to increase adoption of these evidence-based practices
  Interventions: Behavioral: Algorithm
- Control (Active Comparator): Control sites received staff education for pain assessment and management comprised of four one-hour classes
  Interventions: Behavioral: Algorithm

INTERVENTIONS:
Behavioral: Algorithm — The NH pain management algorithm is a series of decision-making tools that begin with regular, comprehensive pain assessment matched to residents' cognitive status and proceed through analgesic therapy appropriate to the character, severity, and pattern of pain.

SUMMARY:
Pain assessment and management deficiencies in nursing homes (NHs) are well documented. Unrelieved pain in this setting results in poorer resident outcomes, including depression, decreased mobility, sleep disturbance, and impaired physical and social functioning. This randomized controlled trial will evaluate the efficacy of a pain management algorithm coupled with intense diffusion strategies in improving pain, physical function and depression among NH residents. Specific aims of the study are to: 1) Evaluate the effectiveness of a pain management algorithm (ALG) coupled with intense diffusion strategies, as compared with pain education (EDU) and weak diffusion strategies, in improving pain, mobility, and depression among NH residents; 2) Determine the extent to which adherence to the ALG and organizational factors are associated with changes in resident outcomes and the extent to which changes in these variables are associated with changes in outcomes; 3) Evaluate the persistence of changes in process and outcome variables at long-term follow-up and 4) Evaluate the relationships among behavioral problems and pain in severely cognitively impaired residents who are unable to provide self-report.

DETAILED DESCRIPTION:
Inadequate pain management in nursing homes (NHs) is well documented. Unrelieved pain in this setting results in depression, decreased mobility, sleep disturbance, and impaired physical and social functioning. This randomized controlled trial will evaluate the efficacy of a pain management algorithm delivered using intense diffusion strategies. Outcomes are facility pain practices and residents' pain, physical function and depression. Specific aims of the study are to: 1) Evaluate the effectiveness of a pain management algorithm (ALG) coupled with intense diffusion strategies, as compared with pain education (EDU) and weak diffusion strategies, in improving pain, mobility, and depression among NH residents; 2) Determine the extent to which adherence to the ALG and organizational factors are associated with changes in resident outcomes and the extent to which changes in these variables are associated with changes in outcomes; 3) Evaluate the persistence of changes in process and outcome variables at long-term follow-up and 4) Evaluate the relationships among behavioral problems and pain in severely cognitively impaired residents who are unable to provide self-report.

ELIGIBILITY:
Inclusion Criteria:

* long-term nursing home residents,
* 65 years and older,
* with moderate or greater pain in the week prior to screening,
* residing in a participating facility,
* who consent to participate (or whose surrogate decisionmaker consents to participation)

Exclusion Criteria:

* short-term stay patients,
* persons less than 65 years,
* residents on hospice

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 396 (Actual)
Dates: Start 2006-09; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain at 3 months | 3 months
  Brief Pain Inventory (self-reporting participants) Nursing Assistant Surrogate Report
Change from Baseline in Pain at 6 months | 6 months post intervention
  Brief Pain Inventory (self-reporting participants) Nursing Assistant Surrogate Report

SECONDARY OUTCOMES:
Change from Baseline in Mobility at 3 months | 3 months
  Functional independence measure - locomotion
Change from Baseline in Agitation at 6 months | 6 months
  Pittsburgh Agitation Scale
Change from Baseline Adherence to Best Practices at 3 months | 3 months
  Pain Management Chart audit Tool; 17 item tool evalauting staff adherence to recommended pain assessment and management practices
Change from Baseline in Depression at 3 months | 3 months
  Cornell Scale for Depression in Dementia
Change from Baseline in Depression at 6 months | 6 months post intervention
  Cornell Scale for Depression in Dementia
Change from Baseline in Mobility at 6 months | 6 months post-intervention
  Functional independence measure - locomotion
Change from Baseline in Adherence to Best Practices at 6 months | 6 months post-intervention
  Pain Management Chart audit Tool; 17 item tool evalauting staff adherence to recommended pain assessment and management practices

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ersek, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Swedish Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Jablonski AM, DuPen AR, Ersek M. The use of algorithms in assessing and managing persistent pain in older adults. Am J Nurs. 2011 Mar;111(3):34-43; quiz 44-5. doi: 10.1097/10.1097/01.NAJ.0000395239.60981.2f. PMID 21346465
- [Background] Ersek M, Polissar N, Neradilek MB. Development of a composite pain measure for persons with advanced dementia: exploratory analyses in self-reporting nursing home residents. J Pain Symptom Manage. 2011 Mar;41(3):566-79. doi: 10.1016/j.jpainsymman.2010.06.009. Epub 2010 Nov 20. PMID 21094018
- [Result] Ersek M, Herr K, Neradilek MB, Buck HG, Black B. Comparing the psychometric properties of the Checklist of Nonverbal Pain Behaviors (CNPI) and the Pain Assessment in Advanced Dementia (PAIN-AD) instruments. Pain Med. 2010 Mar;11(3):395-404. doi: 10.1111/j.1526-4637.2009.00787.x. Epub 2010 Jan 15. PMID 20088854
- [Result] Jablonski A, Ersek M. Nursing home staff adherence to evidence-based pain management practices. J Gerontol Nurs. 2009 Jul;35(7):28-34; quiz 36-7. doi: 10.3928/00989134-20090428-03. PMID 19650621
- [Derived] Ersek M, Neradilek MB, Herr K, Jablonski A, Polissar N, Du Pen A. Pain Management Algorithms for Implementing Best Practices in Nursing Homes: Results of a Randomized Controlled Trial. J Am Med Dir Assoc. 2016 Apr 1;17(4):348-56. doi: 10.1016/j.jamda.2016.01.001. Epub 2016 Feb 17. PMID 26897592
- [Derived] Ersek M, Polissar N, Pen AD, Jablonski A, Herr K, Neradilek MB. Addressing methodological challenges in implementing the nursing home pain management algorithm randomized controlled trial. Clin Trials. 2012 Oct;9(5):634-44. doi: 10.1177/1740774512454243. Epub 2012 Aug 9. PMID 22879574